CLINICAL TRIAL: NCT04110236
Title: Pilot Evaluation of Enhanced Child Adult Relationship Enhancement in Pediatric Primary Care (PriCARE) Intervention
Brief Title: Pilot of Enhanced Child Adult Relationship Enhancement in Pediatric Primary Care
Acronym: PriCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Annie E. Casey Foundation (Other Government); The Pew Charitable Trusts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-016283
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Child Behavior Problem; Parent-Child Relations
Keywords: Child behavior problems; Caregiver child relationship; Primary care
MeSH Terms: interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study team member who will administer the follow-up study interviews will remain blinded to the group status throughout the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immediate PriCARE (Experimental): Caregiver-child dyads assigned to the immediate PriCARE group will receive the PriCARE intervention as soon as possible plus usual treatment. The intervention will last approximately 6-8 weeks. Each group will have approximately 4-13 participants and 1-2 facilitators and will meet 6 times for 1-2 hours per session. Parents are expected to practice the skills they learn with their children between sessions.
  Interventions: Behavioral: PriCARE
- Delayed PriCARE (No Intervention): The delayed PriCARE group will not receive the PriCARE intervention until after their data collection for this study is complete (in 3-6 months). In addition, they will be immediately offered usual treatment. Under usual treatment, patients will be referred to a behavioral health specialist at the discretion of their pediatrician and the office social worker for additional diagnosis and treatment.
- Immediate PriCARE Positive Discipline Module (Experimental): A subset of participants (up to 40 caregiver-child pairs) who were assigned to the immediate PriCARE group will be offered to participate in the PriCARE Positive Discipline Module if they attended at least 4 PriCARE sessions and completed both main study interviews. If they are randomized to the immediate PriCARE Positive Discipline group, they will attend an additional 4-6 sessions 4-6 weeks after completion of the 6-week PriCARE intervention. This module teaches techniques related to behavior reward charts, appropriate timeout protocol, and other positive discipline techniques for handling persistent behaviors not addressed by the other PriCARE skills.
  Interventions: Behavioral: Positive Discipline Module
- Delayed PriCARE Positive Discipline Module (No Intervention): The delayed Positive Discipline group will not receive the Positive Discipline Module intervention until after their third interview data collection is complete (in 2-3 months). In addition, they will be immediately offered usual treatment. Under usual treatment, patients will be referred to a behavioral health specialist at the discretion of their pediatrician and the office social worker for additional diagnosis and treatment.

INTERVENTIONS:
Behavioral: PriCARE — PriCARE is a group caregiver training program designed to improve child behaviors, caregiver-child relationships, parenting capacity, and reduce caregiver stress. Sessions occur in the primary care clinic or virtually. PriCARE uses the 3 P skills (Praise, Paraphrase and Point-out-Behavior). The training starts with skills on giving attention to children's positive, pro-social behaviors, while ignoring minor misbehaviors. The second part of the training teaches skills for giving effective commands in order to set age-appropriate limits and increase compliance. PriCARE includes a stress education section that contextualizes the use of these skills with the types of behaviors and problems exhibited by many children living with psychosocial adversity and familial stress. Caregivers are encouraged to practice the skills with their child in between sessions. Since PriCARE's initial and successful pilot, the intervention has been enhanced in order to increase engagement and effectiveness.
  Other Names: Child Adult Relationship Enhancement in Primary Care
  Arms: Immediate PriCARE
Behavioral: Positive Discipline Module — The PriCARE Positive Discipline Module is a pilot group caregiver training program designed to teach caregivers positive discipline techniques, including appropriate timeout procedures. The sessions are offered in the primary care setting or virtually. This training will supplement the content of the main PriCARE intervention and provide caregivers with skills for addressing difficult behaviors not reduced through positive attention and strategic ignoring. This module will be offered to a subset of CHOP participants who were randomized to the intervention arm, successfully completed the main study interviews, and attended at least 4 out of the 6 PriCARE sessions.
  Other Names: PriCARE Positive Discipline Module
  Arms: Immediate PriCARE Positive Discipline Module

SUMMARY:
The purpose of this study is to evaluate the efficacy of the enhanced PriCARE intervention in improving parenting capacity, decreasing child behavior problems, and reducing risk of child maltreatment at several primary care clinics in Philadelphia and 2 primary care clinics in North Carolina.

DETAILED DESCRIPTION:
Child behavioral concerns are common among families served by Children's Hospital of Philadelphia (CHOP) and University of North Carolina (UNC) pediatric primary care centers. To address this, Child Adult Relationship Enhancement in Pediatric Primary Care (PriCARE) was developed. PriCARE has been evaluated in primary care centers at CHOP and UNC with promising findings with regards to reductions in child behavioral problems. The PriCARE curriculum has now been enhanced with strategies to increase participant engagement, retention of skills, and attendance. Efficacy of this enhanced PriCARE curriculum has not yet been evaluated. Nor has the impact of the PriCARE intervention on child maltreatment risk been explored.

The primary objective of this study is to evaluate the efficacy of the enhanced PriCARE program to improve parenting capacity as measured by the Parenting Scale total score and 3 sub-scales.

The secondary objectives are to:

1. Measure the impact of PriCARE on parent-reported child behavior problems as assessed by the Eyberg Child Behavior Inventory intensity and problems scales.
2. Measure the impact of PriCARE on the quality of the parent-child relationship as measured by the Dyadic Parent-Child Interaction Coding.
3. Measure the impact of PriCARE on the risk of child maltreatment as measured by the Child Abuse Potential Inventory.
4. Identify and describe predictors of attendance in PriCARE groups.
5. Identify and describe modifiers of the efficacy of PriCARE including but not limited to caregiver and child demographics.
6. Assess caregivers' perceptions of the efficacy of PriCARE on improving parenting skills and child behavior as measured by the Therapeutic Attitude Inventory (TAI).
7. Develop and pilot a new PriCARE Positive Discipline Module.
8. Collect pilot data on added benefit of completing the PriCARE Positive Discipline Module.

The investigators will perform a randomized controlled trial (RCT) of the effectiveness of the enhanced PriCARE on objectives listed above among 2- to 6-year-old children and their parents at several CHOP Primary Care Centers and two University of North Carolina primary care sites. The investigators intend to randomize up to 119 child-caregiver pairs (238 subjects) to receive PriCARE immediately plus usual treatment (intervention group) and up to 119 child-parent pairs (238 subjects) to receive PriCARE at a later time plus usual treatment (control group) for a total of up to 238 child-caregiver pairs (476 subjects). All child-caregivers pairs randomized to the control group will be placed on a waitlist and offered PriCARE after completion of data collection. Child maltreatment risk, parenting attitudes and skills, child behavior, and quality of the child-caregiver relationship will be measured at baseline (time 1) and approximately 8-17 weeks after randomization (time 2) for both the intervention and control groups. The follow up interview will also include a brief satisfaction questionnaire for participants randomized to the intervention group. For the subgroup of participants who complete the Positive Discipline Module, these measurements will be repeated approximately 2-4 weeks after completion of the Positive Discipline intervention (time 3).

ELIGIBILITY:
Inclusion Criteria:

* Caregiver is 18 years or older
* Caregiver is English speaking
* Caregiver is legal guardian of child and provides informed consent
* Caregiver has cellular phone with text messaging capacity
* Caregiver is available for scheduled times PriCARE hosts groups
* Child is 2-6 years old
* Caregiver must have the appropriate technological tools and access to participate when in-person sessions are not available
* Child attends one of the CHOP primary care sites in Pennsylvania or one of two University of North Carolina (UNC Children's Primary Care and UNC Pediatrics at Panther Creek) primary care sites

Exclusion Criteria:

* Caregiver has already completed the PriCARE program
* Child has already received a behavioral health diagnosis or is already receiving individualized behavior health therapy or associated medication for Oppositional Defiance Disorder, Conduct Disorder, or Attention- Deficit/Hyperactivity Disorder
* Child is being evaluated for or has been diagnosed with autism
* Child has a cognitive age less than 2 years old as determined by screening questions and/or the referring clinician.
* Child has caused physical injuries, such as bruises or cuts, more than once and on purpose to their caregiver, him/herself, or other children or people

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Change in the Parenting Scale (PS) score from time 1 to time 2 | Baseline (time 1), 8-17 weeks (time 2)
  The primary objective of the study is to evaluate the efficacy of the enhanced PriCARE program to improve parenting capacity as measured by the Parenting Scale (PS), a 30-item questionnaire that assesses dysfunctional parenting discipline strategies. Participants respond to various hypothetical situations with a 7-point Likert scale, where 7 is the "ineffective" end of the scale and a lower overall score indicates more effective parenting. There are 3 scale factors: 1) laxness, 2) over-reactivity, and 3) verbosity. Some items are unrelated to any of these 3 factors. The 11 Laxness items relate to permissive discipline, lack of rule reinforcement and providing positive consequences for misbehaviors. The 10 Over-Reactivity items reflect anger, irritability or meanness. The 7 Verbosity items suggest longer verbal responses such as talking when talking is ineffective. All item responses are averaged to compute the total score. Each factors' items are averaged to compute the factor scores

SECONDARY OUTCOMES:
Change in the Eyberg Child Behavior Inventory (ECBI) score from time 1 to time 2 | Baseline (time 1), 8-17 weeks (time 2)
  The investigators will assess the efficacy of the enhanced PriCARE on decreasing caregiver-reported child behavior problems as measured by the ECBI. The ECBI is a parent rating scale designed to measure conduct problem behaviors in children ages 2-16 years old. The instrument contains 36 items that assess behavior on two scales. The problem scale provides a yes/no problem identification rating for each item, and the sum of yes responses yields a problem score with a potential range from 0 to 36 with a clinical cutoff of 15. The intensity scale provides a frequency-of-occurrence rating for each item, ranging from never (1) to always (7) and the ratings are summed to yield an intensity score with a potential range from 36 to 252 with a clinical cutoff of 131. Higher scores indicate worse outcomes.
Change in the Dyadic Parent-Child Interaction Coding (DPICS) score from time 1 to time 2 | Baseline (time 1), 8-17 weeks (time 2)
  Investigators will assess the efficacy of enhanced PriCARE on impacting the quality of the caregiver-child relationship with the DPICS. Each dyad is observed in 3 standard situations that involve varying levels of parental control and display dyadic interactions targeted by PriCARE: child-led play, caregiver-led play, clean-up. The coding manual has definitions, examples, and guidelines for deciding how to code the 24 standard caregiver and child behaviors. The interactions are video-recorded and coded by a blinded research assistant. Zero, or not observed, is the minimum for all behaviors. The total score is the sum of the coded behaviors within each category, thus there is no set maximum. A second research assistant re-codes 25% of randomly selected videos to check for coding reliability. Reliability will be assessed using % agreement, intraclass correlations, and Cohen's kappa. Comparing pre- and post-intervention videos will demonstrate caregiver and child behavior changes.
Change in the Child Abuse Potential Inventory (CAPI) score from time 1 to time 2 | Baseline (time 1), 8-17 weeks (time 2)
  CAPI change scores from time 1 to time 2 will be measured. CAPI, a 160-item survey, measures traits & parenting styles typical of known physical child abusers. Each item has a weighted value based on if agree vs. disagree is chosen and then the values are summed. Child physical abuse scores range from 0-486 with higher scores indicating caregiver has traits similar to those of known child abusers and has a higher risk of abuse. Ranges for factor scales are: distress (0-261), rigidity (0-64), unhappiness (0-69), problems with child and self (0-30), problems with family (0-38), problems with others (0-24) Higher factor scores imply higher symptom levels. Three validity scales and ranges are: lie (0-18), random (0-18), inconsistency (0-20). Ego-strength score ranges from 0-40 with higher score indicating more emotional stability. Loneliness score ranges from 0-15; higher score means more isolation.
Therapeutic Attitudes Inventory (TAI) | 8-17 weeks (time 2)
  The investigators will assess caregivers' perceptions of the efficacy of PriCARE on improving parenting skills and child behavior as measured by the TAI. The TAI is a brief 10-question satisfaction measure of parent training and parent-child treatments. Questions are answered on a 5-point Likert scale with 1 indicating the lowest ("nothing", "much worse than before", "much less confident", etc.) and 5 indicating the highest ("very many useful techniques", "very much better than before", "more confident", etc.). Responses are added together and greater TAI total scores indicate greater levels of participant satisfaction. The potential scores range from 10-50.

OTHER OUTCOMES:
Change in the Parenting Scale (PS) score from time 2 to time 3 | 8-17 weeks (time 2) to 16-30 weeks (time 3)
  Change in PS from time 2 to time 3 will be measured in the subset of CHOP participants completing the Positive Discipline Module. PS is a 30-item questionnaire that assesses dysfunctional parenting discipline strategies. Participants respond to various hypothetical situations with a 7-point Likert scale, where 7 is the "ineffective" end of the scale and a lower overall score indicates more effective parenting. There are 3 scale factors: 1) laxness, 2) over-reactivity, and 3) verbosity. Some items are unrelated to any of these 3 factors. The 11 Laxness items relate to permissive discipline, lack of rule reinforcement and providing positive consequences for misbehaviors. The 10 Over-Reactivity items reflect anger, irritability or meanness. The 7 Verbosity items suggest longer verbal responses such as talking when talking is ineffective. All item responses are averaged to compute the total score. Each factors' items are averaged to compute the factor scores.
Change in the Eyberg Child Behavior Inventory (ECBI) score from time 2 to time 3 | 8-17 weeks (time 2), 16-30 weeks (time 3)
  Change in ECBI scores from time 2 to time 3 will be measured in the subset of CHOP participants completing the Positive Discipline Module. The ECBI is a parent rating scale designed to measure conduct problem behaviors in children ages 2-16 years old. The instrument contains 36 items that assess behavior on two scales. The problem scale provides a yes/no problem identification rating for each item, and the sum of yes responses yields a problem score with a potential range from 0 to 36 with a clinical cutoff of 15. The intensity scale provides a frequency-of-occurrence rating for each item, ranging from never (1) to always (7) and the ratings are summed to yield an intensity score with a potential range from 36 to 252 with a clinical cutoff of 131. Higher scores indicate worse outcomes.
Change in the Dyadic Parent-Child Interaction Coding (DPICS) score from time 2 to time 3 | 8-17 weeks (time 2), 16-30 weeks (time 3)
  Change in DPICS scores from time 2 to time 3 will be measured in the subset of CHOP participants completing the Positive Discipline Module. Each dyad is observed in 3 standard situations that involve varying levels of parental control and display dyadic interactions targeted by PriCARE: child-led play, caregiver-led play, clean-up. The coding manual has definitions, examples, and guidelines for deciding how to code the 24 standard caregiver and child behaviors. The interactions are video-recorded and coded by a blinded research assistant. Zero, or not observed, is the minimum for all behaviors. The total score is the sum of the coded behaviors within each category, thus there is no set maximum. A second research assistant re-codes 25% of randomly selected videos to check for coding reliability. Reliability will be assessed using % agreement, intraclass correlations, and Cohen's kappa. Comparing pre- and post-intervention videos will demonstrate caregiver and child behavior changes.
Therapeutic Attitudes Inventory (TAI) at time 3 | 16-30 weeks (time 3)
  The investigators will assess caregivers' perceptions of the efficacy of PriCARE on improving parenting skills and child behavior as measured by the TAI at time 3 for the subset of participants completing the Positive Discipline Module. The TAI is a brief 10-question satisfaction measure of parent training and parent-child treatments. Questions are answered on a 5-point Likert scale with 1 indicating the lowest ("nothing", "much worse than before", "much less confident", etc.) and 5 indicating the highest ("very many useful techniques", "very much better than before", "more confident", etc.). Responses are added together and greater TAI total scores indicate greater levels of participant satisfaction. The potential scores range from 10-50.
Change in the Child Abuse Potential Inventory (CAPI) score from baseline to time 2 to time 3 | 8-17 weeks (time 2), 16-30 weeks (time 3)
  CAPI change scores from time 2 to 3 will be measured in subjects participating in the Positive Discipline Module. CAPI, a 160-item survey, measures traits & parenting styles typical of known physical child abusers. Each item has a weighted value based on if agree vs. disagree is chosen and then the values are summed. Child physical abuse scores range from 0-486 with higher scores indicating the caregiver has traits similar to those of known child abusers and has a higher risk of abuse. Ranges for factor scales are: distress (0-261), rigidity (0-64), unhappiness (0-69), problems with child and self (0-30), problems with family (0-38), problems with others (0-24) Higher factor scores imply higher symptom levels. Three validity scales and ranges are: lie (0-18), random (0-18), inconsistency (0-20). Ego-strength score ranges from 0-40 with higher score indicating more emotional stability. Loneliness score ranges from 0-15; higher score means more isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Wood, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weitzman C, Wegner L; Section on Developmental and Behavioral Pediatrics; Committee on Psychosocial Aspects of Child and Family Health; Council on Early Childhood; Society for Developmental and Behavioral Pediatrics; American Academy of Pediatrics. Promoting optimal development: screening for behavioral and emotional problems. Pediatrics. 2015 Feb;135(2):384-95. doi: 10.1542/peds.2014-3716. PMID 25624375
- [Background] Bultas MW, McMillin SE, Broom MA, Zand DH. Brief, Rapid Response, Parenting Interventions Within Primary Care Settings. J Behav Health Serv Res. 2017 Oct;44(4):695-699. doi: 10.1007/s11414-015-9479-2. PMID 26289564
- [Background] Querido JG, Warner TD, Eyberg SM. Parenting styles and child behavior in African American families of preschool children. J Clin Child Adolesc Psychol. 2002 Jun;31(2):272-7. doi: 10.1207/S15374424JCCP3102_12. PMID 12056110
- [Background] Asarnow JR, Rozenman M, Wiblin J, Zeltzer L. Integrated Medical-Behavioral Care Compared With Usual Primary Care for Child and Adolescent Behavioral Health: A Meta-analysis. JAMA Pediatr. 2015 Oct;169(10):929-37. doi: 10.1001/jamapediatrics.2015.1141. PMID 26259143
- [Background] Meadows T, Valleley R, Haack MK, Thorson R, Evans J. Physician "costs" in providing behavioral health in primary care. Clin Pediatr (Phila). 2011 May;50(5):447-55. doi: 10.1177/0009922810390676. Epub 2010 Dec 30. PMID 21196418
- [Background] Ward-Zimmerman B, Cannata E. Partnering with pediatric primary care: Lessons learned through collaborative colocation. Professional Psychology: Research and Practice. 2012;43(6):596-605.
- [Background] Schuhmann EM, Foote RC, Eyberg SM, Boggs SR, Algina J. Efficacy of parent-child interaction therapy: interim report of a randomized trial with short-term maintenance. J Clin Child Psychol. 1998 Mar;27(1):34-45. doi: 10.1207/s15374424jccp2701_4. PMID 9561935
- [Background] Eyberg SM, Ross AW. Assessment of Child Behavior Problems: The Validation of a New Inventory. J Clin Child Psycho. 1978.
- [Background] McKelvey LM, Burrow NA, Balamurugan A, Whiteside-Mansell L, Plummer P. Effects of home visiting on adolescent mothers' parenting attitudes. Am J Public Health. 2012 Oct;102(10):1860-2. doi: 10.2105/AJPH.2012.300934. Epub 2012 Aug 16. PMID 22897545
- [Background] Arnold DS, O'Leary SG, Wolff LS, Acker MM. The Parenting Scale: A measure of dysfunctional parenting in discipline situations. Psychological Assessment. 1993;5(2):137-44. doi: 10.1037/1040-3590.5.2.137.
- [Background] Karazsia B, Dulmen M, Wildman B. Confirmatory Factor Analysis of Arnold et al.'s Parenting Scale Across Race, Age, and Sex. Journal of Child & Family Studies. 2008;17(4):500-16. doi: 10.1007/s10826-007-9170-1. PubMed PMID: 32587293.
- [Background] Steele RG, Nesbitt-Daly JS, Daniel RC, Forehand R. Factor Structure of the Parenting Scale in a Low-Income African American Sample. Journal of Child & Family Studies. 2005;14(4):535-49. doi: 10.1007/s10826-005-7187-x. PubMed PMID: 18485834.
- [Background] Irvine AB, Biglan A, Smolkowski K, Ary DV. The value of the Parenting Scale for measuring the discipline practices of parents of middle school children. Behav Res Ther. 1999 Feb;37(2):127-42. doi: 10.1016/s0005-7967(98)00114-4. PMID 9990744
- [Background] Burns G, Patterson D. Conduct problem behaviors in a stratified random sample of children and adolescents: New Standardization data on the Eyberg Child Behavior Inventory. Psychological Assessment. 1990;2:291-297.
- [Background] Colvin A, Eyberg S, Adams C. Restandardization of the Eyberg Child Behavior Inventory. 1999
- [Background] Robinson E, Eyberg S, Ross W. The standardization of an inventory of child conduct problem behaviors. Journal of Clinical Child Psychology. 1980;9:22-28.
- [Background] Funderburk B, Eyberg SM, Rich BA, Behar L. Further Psychometric Evaluation of the Eyberg and Behar Rating Scales for Parents and Teachers of Preschoolers. Early Education and Development. 2003;14(1):67-81.
- [Background] Webster-Stratton C, Reid MJ, Hammond M. Treating children with early-onset conduct problems: intervention outcomes for parent, child, and teacher training. J Clin Child Adolesc Psychol. 2004 Mar;33(1):105-24. doi: 10.1207/S15374424JCCP3301_11. PMID 15028546
- [Background] Achenbach T. Integrative Guide to the 1991 CBCL/4-18, YSR, and TRF Profiles. Burlington, VT: University of Vermontm 1991.
- [Background] Eyberg S, Pincus D. Eyberg Child Behavior Inventory and Stutter-Eyberg Student Behavior Inventory-revised: Professional manual. Odessa, FL1999.
- [Background] Brestan EV JJ, Rayfield AD, Eybert SM. A consumer satisfaction measure for parent-child treatments and its relation to measures of child behavior change. Behavior Therapy. 1999;30:17-30.
- [Background] Eyberg S, Bessmer J, Newcomb K, Edwards D, Robinson E. Dyadic Parent-Child Interaction Coding Scheme II: A manual. Unpublished manuscript, University of Florida. 1994.
- [Background] Eyberg SM, Nelson MM, Duke M, Boggs SR. Manual for the Dyadic Parent-Child Interaction Coding System Third Edition. 2004.
- [Background] Robinson EA, Eyberg SM. The dyadic parent-child interaction coding system: standardization and validation. J Consult Clin Psychol. 1981 Apr;49(2):245-50. doi: 10.1037//0022-006x.49.2.245. No abstract available. PMID 7217491
- [Background] Bessmer JL. The Dyadic Parent-Child Interaction Coding System II (DPICS II): Reliability and validity, ProQuest Information & Learning; 1998.
- [Background] Foote RC. The Dyadic Parent-Child Interaction Coding System II (DPICS II): Reliability and validity with father-child dyads, ProQuest Information & Learning; 2000.
- [Background] Webster-Stratton C. Comparisons of behavior transactions between conduct-disordered children and their mothers in the clinic and at home. J Abnorm Child Psychol. 1985 Jun;13(2):169-83. doi: 10.1007/BF00910640. PMID 4008751
- [Background] Webster-Stratton C. Advancing videotape parent training: a comparison study. J Consult Clin Psychol. 1994 Jun;62(3):583-93. doi: 10.1037//0022-006x.62.3.583. PMID 8063985
- [Background] Webster-Stratton C. Preventing conduct problems in Head Start children: strengthening parenting competencies. J Consult Clin Psychol. 1998 Oct;66(5):715-30. doi: 10.1037//0022-006x.66.5.715. PMID 9803690
- [Background] Milner J. The Child Abuse Potential Inventory: Manual. 2nd ed ed. Webster, NC: Psytec; 1986.
- [Background] Milner J. An interpretive manual for the Child Abuse Potential Inventory. DeKalb, IL: Psytec; 2006.
- [Background] Milner JS. Assessing physical child abuse risk: The Child Abuse Potential Inventory. Clinical Psychology Review. 1994;14:547-583.
- [Background] Begle AM, Dumas JE, Hanson RF. Predicting child abuse potential: an empirical investigation of two theoretical frameworks. J Clin Child Adolesc Psychol. 2010;39(2):208-19. doi: 10.1080/15374410903532650. PMID 20390812
- [Derived] Kiely J, DePaul E, Rojas S, Cortes S, Schilling S, Dougherty S, Wood JN. Evaluation of Virtual Enhanced Child Adult Relationship Enhancement in Primary Care Intervention. J Dev Behav Pediatr. 2024 Sep-Oct 01;45(5):e439-e447. doi: 10.1097/DBP.0000000000001292. Epub 2024 Jun 21. PMID 39413305